CLINICAL TRIAL: NCT04997278
Title: Coordinated Reset Spinal Cord Stimulation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jaimie M. Henderson, Professor of Neurosurgery, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 44884
Record Dates: First submitted 2021-07-12; First posted 2021-08-09 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Pain, Neuropathic; Failed Back Surgery Syndrome
Keywords: spinal cord stimulation; chronic pain; neuropathic pain; failed back surgery syndrome
MeSH Terms: conditions — Neuralgia; Failed Back Surgery Syndrome; Chronic Pain

STUDY DESIGN:
Intervention Model Description: A single group will be studied, comparing the new stimulation paradigm with the standard paradigm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Coordinated Reset- Spinal Cord Stimulation (Experimental): All subjects will undergo spinal cord stimulation (SCS) implantation and will be optimized on standard SCS (sSCS) settings using the standard clinical protocol, including paresthesia mapping, threshold finding, and adjustment of stimulation parameters to provide reduction in pain. Therapeutic sSCS will be maintained for a minimum of one month prior to baseline assessment. Following a washout period of three hours assessments will be performed and Coordinated Reset- spinal cord stimulation (CR-SCS) will be enabled by means of a firmware upgrade. Personnel from Boston Scientific will perform this upgrade. The simulator will then be programmed to deliver CR-SCS. At the end of one month of CR-SCS (with stimulation parameters similarly held constant for the last 7 days), baseline assessment will be repeated after a three hour washout period. Finally, a firmware downgrade will be performed by Boston Scientific Personnel, and patients will be treated with sSCS at their previous settings.
  Interventions: Device: Coordinated Reset spinal cord stimulation

INTERVENTIONS:
Device: Coordinated Reset spinal cord stimulation — Abnormal neuronal synchrony in terms of enhanced 4-9 Hz theta oscillations in EEG/MEG recordings appears to be an important pathophysiological finding in patients with neurogenic pain. To specifically counteract abnormal neuronal synchrony, we here set out to perform Coordinated Reset (CR)-Spinal Cord Stimulation (SCS). CR stimulation (Tass, 2003) aims at an anti-kindling, i.e. an "unlearning" or resetting of abnormal neuronal synchrony and abnormal synaptic connectivity, and, hence, long-lasting, sustained therapeutic effects that persist following cessation of stimulation (Tass & Majtanik, 2006).

SUMMARY:
The goal of this study is to evaluate whether a new spinal cord stimulation paradigm, called Coordinate Reset (CR) Stimulation, can provide equivalent or better pain relief with reduced energy requirements. The investigators will test this new stimulation paradigm in patients who are already undergoing spinal cord stimulation surgery. The investigators will also study whether there are changes in electroencephalography (brain waves) associated with this new stimulation paradigm.

The investigators hope to learn whether CR stimulation can provide equivalent or better pain relief with reduced energy requirements. They also hope to learn whether there are changes in brain function with effective CR stimulation compared to conventional stimulation.

This study will be testing a specific stimulation paradigm in people who have already consented to have spinal cord stimulation performed for treatment of their chronic pain.

DETAILED DESCRIPTION:
Study subjects will be identified from the pool of candidates for spinal cord stimulation (SCS) therapy at Stanford University. Subjects will have undergone a successful trial of Boston Scientific spinal cord stimulation and will either be candidates for permanent stimulator implantation, or will have already undergone implantation. Ten subjects will be recruited over a one year period.

Following informed consent, subjects will be assessed to assure that they meet the criteria for study entry. All subjects will undergo SCS implantation and will be optimized on standard SCS (sSCS) settings using the standard clinical protocol, including paresthesia mapping, threshold finding, and adjustment of stimulation parameters to provide reduction in pain. Therapeutic sSCS will be maintained for a minimum of one month prior to baseline assessment.

Baseline assessments will be conducted following discontinuation of SCS for 24 hours. This assessment battery includes a physical and neurological exam, visual analog scale (VAS) score, Oswestry Disability Index, SF-12 and Global Assessment of Functioning, as well as EEG recordings (spontaneous EEG recording + dedicated pain-related evoked response recording). Following this baseline assessment, sSCS will be delivered for one month. Stimulation parameters will be held constant for the last 7 days of this period. During this time, subjects will use the CamNtech Pro-Diary wrist-worn data entry system to rate their back pain, leg pain and overall pain (3 questions), 3 times per day (morning, afternoon evening). The Pro-Diary allows for configurable, portable data entry as well as actigraphy.

The full assessment battery will be repeated, and the stimulator deactivated.

Following a washout period of three hours, VAS and EEG recordings will be performed. CR-SCS will be enabled by means of a firmware upgrade. Personnel from Boston Scientific will perform this upgrade. The stimulator will then be programmed to deliver CR-SCS. At the end of one month of CR-SCS (with stimulation parameters similarly held constant for the last 7 days), the assessment battery will be repeated, and VAS and EEG recordings will again be performed after a three hour washout period. Finally, a firmware downgrade will be performed by Boston Scientific Personnel, and patients will be treated with sSCS at their previous settings.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic neuropathic lower extremity pain, without back pain, who have consented to undergo or are undergoing spinal cord stimulation (SCS)
2. Age 22 to 70
3. Fluent in English and able to independently provide consent
4. Patients treated with conventional SCS for at least 3 months prior to commencement of study, either newly implanted or already implanted.
5. Patients have pronounced pain, i.e. visual analog scale score (VAS) ≥6 and respond to conventional SCS, i.e. VAS reduction of at least 50% with SCS.

Exclusion Criteria:

1. Significant psychiatric problems, including unrelated clinically significant depression as determined by the investigator.
2. Current drug or alcohol abuse as determined by the investigator.
3. Any history of recurrent or unprovoked seizures.
4. Any significant medical condition that is likely to interfere with study procedures or likely to confound evaluation of study endpoints, including any terminal illness with survival <12 months.
5. Females who are pregnant, breastfeeding, or are of childbearing potential and planning to get pregnant during the course of the study or not using adequate contraception
6. On anticoagulation therapy

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Pain relief | One month
  Difference in mean reduction in visual analog scale (VAS) score between sSCS and CR-SCS for leg pain and / or back pain compared to baseline, with 0 indicating no pain and 100 indicating worst pain.

SECONDARY OUTCOMES:
Activity level | One month
  Use of CamNtech Pro-Diary wrist-worn data entry system to rate back pain, leg pain and overall pain (3 questions), 3 times per day (morning, afternoon evening). Patients will rate their pain on a 0-10 Visual Analog scale with 0 indicating no pain and 100 worst pain.
Oswestry Disability Index, Sort Form-12 | One month
  Oswestry Disability Index, Sort From-12 (also known as the Oswestry Low Back Pain Disability Questionnaire) is a 12 item short survey that measure a patient's permanent functional disability. Each section is scored on a 0-5 scale, 5 representing the greatest disability.
Global Assessment of functioning Scale (GAF) | One month
  The Global Assessment of Functioning (GAF) scale is used to rate how serious a mental illness may be. It measures how much a person's symptoms affect their day-to-day life on a scale of 0 to 100, with higher scores indicating that the subject is better at handling daily activities.
Electroencephalography (EEG) | One month
  EEG activity will be quantified by means theta power (4-9 Hz), with decreases in theta power related to decreased pain. Theta power will be measured pre and post treatment.
Event Related Potentials (ERP) | One month
  During the EEG, we will analyzed ERPs in response to each stimuli during stimulation. Changes in amplitude (micro-volts) will be analyzed pre and post treatment. ERP activity is exploratory.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Health Care, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
No IPD shared outside of Stanford